CLINICAL TRIAL: NCT06303960
Title: The Comparison of Treatment Results Between Cerebellar DBS and Vagus Stimulation for Post-stroke Motor Rehabilitation: a Randomized Clinical Trial
Brief Title: Cerebellar Deep Brain Stimulation or VNS for Chronic Post-stroke Motor Rehabilitation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VNS or DBS for stroke
Record Dates: First submitted 2024-02-05; First posted 2024-03-12 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Hemiparesis; Cerebellar Deep Brain Stimulation; VNS; Limb Motor Function Rehabilitation
MeSH Terms: conditions — Stroke; Paresis | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bilateral Cerebellar deep brain stimulation (Active Comparator): Following enrollment, participants underwent 1 month of upper-extremity rehabilitation twice per week to rule out potential for recovery with rehabilitation therapy alone. Thereafter, each participant underwent surgical implantation of the DBS system, with the lead implanted in the DN contralateral to the stroke-affected cerebral hemisphere. 1 months later, DBS was activated bilaterally.
  Interventions: Device: Bilateral Cerebellar deep brain stimulation
- Unilateral Cerebellar deep brain stimulation (Active Comparator): Following enrollment, participants underwent 1 month of upper-extremity rehabilitation twice per week to rule out potential for recovery with rehabilitation therapy alone. Thereafter, each participant underwent surgical implantation of the DBS system, with the lead implanted in the DN contralateral to the stroke-affected cerebral hemisphere. 1 months later, DBS was activated unilaterally.
  Interventions: Device: Unilateral Cerebellar deep brain stimulation
- Vagus Nerve Stimulation (Experimental): Following enrollment, participants underwent 1 month of upper-extremity rehabilitation twice per week to rule out potential for recovery with rehabilitation therapy alone. Thereafter, each participant underwent surgical implantation of the VNS system. 1 months later, VNS was activated unilaterally.
  Interventions: Device: Vagus Nerve Stimulation

INTERVENTIONS:
Device: Bilateral Cerebellar deep brain stimulation — Participants underwent stereotactic implantation of a single DBS lead in the area of the cerebellar DN contralateral to the lesioned cerebral hemisphere using a frame-based technique similar to that used in DBS for movement disorders. All participants received an 4-channel lead (Medtronic,3389）with electrode arrays up to 15.5 mm in length. Then bilateral stimulation was activated after 1 month post-DBS
  Arms: Bilateral Cerebellar deep brain stimulation
Device: Unilateral Cerebellar deep brain stimulation — Participants underwent stereotactic implantation of a single DBS lead in the area of the cerebellar DN contralateral to the lesioned cerebral hemisphere using a frame-based technique similar to that used in DBS for movement disorders. All participants received an 4-channel lead (Medtronic,3389）with electrode arrays up to 15.5 mm in length. Then unilateral stimulation was activated after 1 month post-DBS
  Arms: Unilateral Cerebellar deep brain stimulation
Device: Vagus Nerve Stimulation — Device implantation was done under general anaesthesia. A horizontal neck crease incision was created left of the midline at the level of the cricoid cartilage. After the vagus nerve was identified, the stimulation lead was wrapped around the vagus nerve. The lead was then tunnelled subcutaneously to the pulse generator device which was contained in a subcutaneous pocket in the pectoral region.
  Arms: Vagus Nerve Stimulation

SUMMARY:
Upper-extremity impairment after stroke remains a major therapeutic challenge and a target of neuromodulation treatment efforts.In this open-label, randomized phase I trial, we applied deep brain stimulation to the cerebellar dentate nucleus combined with bilateral or unilateral stimulation. Vagus nerve stimulation was also conducted for motor function after ischaemic Stroke.We hypothesized that cerebellar stimulation was superior to vagus stimulation as the motor rehabilitation after stroke benefits from both side of cerebellum.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals suffered a first-time, unilateral, ischemic stroke in the middle cerebral artery territory that spared the diencephalon and basal ganglia 12-36 months before surgery.
* Individuals with persistent moderate-to-severe upper-extremity hemiparesis as defined by an FM-UE score of ≤42
* Sufficient upper-extremity motor ability to engage in rehabilitation (that is, a score of ≥1 on the FM-UE elbow flexion, elbow extension or finger mass flexion or extension).

Exclusion Criteria:

* Excessive spasticity or contracture of the upper-extremity muscles (that is, Modified Ashworth Scale = 4)
* Severe cognitive impairment (Mini Mental State Examination < 24)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-06-07 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
FM-UE scores between cerebellar DBS and VNS | 12 months after device implantation
  The outcomes includes each participant's Fugl-Meyer assessment scale (FM-UE) scores for each monthly visit. FM-UE scores range from 0 to 100 and the higher scores indicated better outcome of movement.

SECONDARY OUTCOMES:
Arm Motor Ability Test (AMAT) between cerebellar DBS and VNS | 12 months after device implantation
  The outcomes includes each participant's the Arm Motor Ability Test (AMAT) for each monthly visit. AMAT scores range from 0 to 57 and the higher scores indicated better outcome of movement.
the Nine-Hole Peg Test between cerebellar DBS and VNS | 12 months after device implantation
  The outcomes includes each participant's the Nine-Hole Peg Test for each monthly visit.
the Bilateral Box and Block Test between cerebellar DBS and VNS | 12 months after device implantation
  The outcomes includes each participant's the Bilateral Box and Block Test for each monthly visit.
Short Form Health Survey (SF-12) between cerebellar DBS and VNS | 12 months after device implantation
  The outcomes includes each participant's score of Short Form Health Survey (SF-12) for each monthly visit. SF-12 scores range from 0 to 60 and the higher scores indicated better outcome of movement.
the EuroQol Five Dimensions Questionnaire (EQ-5D) between cerebellar DBS and VNS | 12 months after device implantation
  The outcomes includes each participant's score of the EuroQol (EQ-5D) scores range from 0 to 36 for each monthly visit.
the Beck Depression Inventory or the Beck Anxiety Inventory between cerebellar DBS and VNS | 12 months after device implantation
  The outcomes includes each participant's score of the Beck Depression Inventory or the Beck Anxiety Inventory for each monthly visit.
nerve conduction velocity between cerebellar DBS and VNS | 12 months after device implantation
  The outcomes includes each participant's nerve conduction velocity for each monthly visit recorded by flexible electrode.
safety and feasibility of VNS and cerebellar DBS | 12 months after device implantation
  The incidence of adverse events including hemorrhages, infections, deaths or major perioperative complications during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Chao Zhang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) could be available to other researchers by request of email